CLINICAL TRIAL: NCT04012996
Title: A Multi-Center, Prospective, Randomized Controlled Trial Comparing the Safety and Effectiveness of Prodisc® C SK and Prodisc® C Vivo to Mobi-C® Cervical Disc in the Treatment of Two-Level Symptomatic Cervical Disc Disease (SCDD)
Brief Title: 2-level Cervical Disc Replacement Comparing Prodisc C SK & Vivo to Mobi-C
Acronym: SMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centinel Spine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAL-P-0022
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Symptomatic Cervical Disc Disease
Keywords: symptomatic cervical disc disease; SCDD; neck pain; radiculopathy; myelopathy; cervical spine pain; neck surgery; cervical surgery; arm numbness; hand numbness; arm tingling; hand tingling; arm weakness
MeSH Terms: conditions — Neck Pain; Radiculopathy; Spinal Cord Diseases; Paresis

STUDY DESIGN:
Intervention Model Description: multi-center, prospective, randomized, controlled comparison
Who Masked: Participant
Masking Description: Patient is blinded to their treatment randomization until after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational (Experimental): Two-level prodisc C SK and/or prodisc C Vivo
  Interventions: Device: prodisc C SK and/or Vivo
- Control (Active Comparator): Two-level Mobi-C device
  Interventions: Device: Mobi-C Cervical Disc

INTERVENTIONS:
Device: prodisc C SK and/or Vivo — Subjects will be randomized in a 2:1 ratio either to the two-level prodisc C SK or prodisc C Vivo device (investigational group) or to the two-level Mobi-C device (control group).
  Arms: Investigational
Device: Mobi-C Cervical Disc — Subjects will be randomized in a 2:1 ratio either to the two-level prodisc C SK or prodisc C Vivo device (investigational group) or to the two-level Mobi-C device (control group).
  Arms: Control

SUMMARY:
A multi-center, prospective, randomized, controlled comparison of the prodisc C SK and prodisc C Vivo to the control, a similar, legally marketed total disc replacement device in subjects with symptomatic cervical disc disease (SCDD).

DETAILED DESCRIPTION:
The clinical trial is to demonstrate that prodisc C SK and prodisc C Vivo are at least as safe and effective as a similar, currently marketed cervical disc prosthesis to treat symptomatic cervical disc disease (SCDD) in subjects at two contiguous levels from C3 to C7 who are unresponsive to conservative management. Subjects will be randomized in a 2:1 ratio to either the two-level prodisc C SK or prodisc C Vivo device (investigational group) or to the two-level Mobi-C device (control group). Subjects will be followed for at least 2 years and up to 5 years. Subjects will be required to complete subject questionnaires, have X-rays and undergo neurological assessments during the follow up visits as specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤69 years.
2. Diagnosis of radiculopathy or myelopathy with radiculopathy of the cervical spine, with pain, paresthesias or paralysis in a specific nerve root distribution C3 through C7, including at least one of the following:
3. Symptomatic cervical disc disease (SCDD) at two contiguous levels from C3 to C7.
4. Radiographically determined pathology at the level to be treated correlating to primary symptoms.
5. Unresponsive to non-operative, conservative treatment (rest, heat, electrotherapy, physical therapy, chiropractic care and/or analgesics)

Exclusion Criteria:

1. Have more than one immobile vertebral level between C1 to C7 from any cause including but not limited to congenital abnormalities and osteoarthritic "spontaneous" fusions.
2. Have previous trauma to the C3 to C7 levels resulting in significant bony or disco-ligamentous cervical spine injury.
3. Have had a prior cervical TDR or fusion procedure at any level.
4. Have osteoporosis or is at increased risk of osteoporosis
5. Have active malignancy that included a history of any invasive malignancy (except non-melanoma skin cancer), unless the subject had been treated with curative intent and there had been no clinical signs or symptoms of the malignancy for at least 5 years.
6. Have known allergies to cobalt, chromium, molybdenum, titanium, nickel or polyethylene.
7. Have rheumatoid arthritis, lupus, or other autoimmune disease that affect the musculoskeletal system.
8. Have concomitant conditions requiring daily, high-dose oral and/or inhaled steroids.
9. Have a Body Mass Index (BMI) > 40 kg/m2.
10. Taking medications known to potentially interfere with bone/soft tissue healing (e.g., high-dose oral and/or inhaled steroids, immunosuppressant medication, chemotherapeutic agents).
11. Have a current history of heavy smoking (more than one pack of cigarettes per day).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2028-05-13 (Estimated)

PRIMARY OUTCOMES:
Composite clinical success rate of the two-level prodisc C SK and prodisc C Vivo will be no worse than marketed cervical disc prosthesis (Mobi-C) | 24 months
  Includes assessments such as NDI and neurological improvement.

CONTACTS AND LOCATIONS:
Overall Officials: James Kuras, Study Director — Centinel Spine
Locations (30):
- United States (30):
  - Flagstaff Bone and Joint, Flagstaff, Arizona
  - Todd Lanman, MD, Inc., Beverly Hills, California
  - Doctors Outpatient Center for Surgery, Los Angeles, California
  - Sutter Health - Palo Alto Medical Foundation, Palo Alto, California
  - Sutter Health, Sacramento, California
  - HCA Healthcare, Lone Tree, Colorado
  - Sky Ridge Medical Center Campus, Lone Tree, Colorado
  - Center for Spine and Orthopedics, Scientific Education and Research Foundation, Thornton, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - St. Vincent's Neurosurgery, Jacksonville, Florida
  - Kennedy-White Orthopaedic Center, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Florida Orthopaedic Institute, Temple Terrace, Florida
  - Indiana Spine Group, Carmel, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - University Spine Center, Wayne, New Jersey
  - NYU Langone Orthopedic Hospital, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Northwell Health, Lenox Hill Hospital, New York, New York
  - Axis Neurosurgery and Spine, Williamsville, New York
  - M3-Emerging Medical Resarch, Durham, North Carolina
  - SVCMC Solon Medical - Northern Ohio Surgery Center, Beachwood, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - DFW Center for Spinal Disorders, Fort Worth, Texas
  - Texas Back Institute, Plano, Texas
  - Texas Spine Care Center, San Antonio, Texas
  - The Disc Replacement Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No